CLINICAL TRIAL: NCT00310804
Title: A Phase III, Randomized, Controlled, Observer-Blind, Multi-Center Study to Evaluate Safety, Tolerability and Immunogenicity of a Single Intramuscular Dose of Three Lots of a Trivalent Subunit Influenza Vaccine Produced in Mammalian Cell Culture Or of a Trivalent Subunit Influenza Vaccine Produced in Embryonated Hen Eggs, in Healthy Adult Subjects Aged >=18 to <=60
Brief Title: Safety and Immunogenicity of 3 Lots of Cell-derived Subunit Influenza Vaccine as Compared to 1 Lot to Egg-derived Subunit Influenza Vaccine in Healthy Adults (>=18 to <=60)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P9; EUDRACT: 2005-002257-47
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Influenza
Keywords: Influenza; Flu; Cell-Derived; Egg-Derived; Healthy Adults; Safety; Immunogenicity; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- cTIV_lot 1 (Experimental)
  Interventions: Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 1 (cTIV)
- cTIV_lot 2 (Experimental)
  Interventions: Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 2 (cTIV)
- cTIV_lot 3 (Experimental)
  Interventions: Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 3 (cTIV)
- TIV group (Active Comparator)
  Interventions: Biological: Egg-Derived Trivalent Subunit Influenza Vaccine (TIV)

INTERVENTIONS:
Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 1 (cTIV) — One single 0.5ml intramuscular injection of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 1
  Arms: cTIV_lot 1
Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 2 (cTIV) — One single 0.5ml intramuscular injection of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 2
  Arms: cTIV_lot 2
Biological: Cell-Derived Trivalent Subunit Influenza Vaccine Lot 3 (cTIV) — One single 0.5ml intramuscular injection of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 3
  Arms: cTIV_lot 3
Biological: Egg-Derived Trivalent Subunit Influenza Vaccine (TIV) — One single 0.5ml intramuscular injection of Egg Derived Trivalent Subunit Influenza Vaccine (TIV).
  Arms: TIV group

SUMMARY:
The present study aims to evaluate safety, tolerability and immunogenicity of three lots of Chiron's cell-derived subunit influenza vaccine in healthy adult subjects as compared to a conventional egg-derived control vaccine licensed in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to <61 years of age
2. mentally competent to understand the nature, the scope and the consequences of the study
3. able and willing to give written informed consent prior to study entry
4. in good health as determined by:

   1. medical history,
   2. physical examination,
   3. clinical judgment of the Investigator.

Exclusion Criteria:

1. unwilling or unable to give written informed consent to participate in the study
2. participation in another clinical trial of an investigational agent within 90 days prior to Visit 1 and throughout the entire study
3. currently experiencing an acute infectious disease
4. any serious disease, such as, for example:

   1. cancer,
   2. autoimmune disease (including rheumatoid arthritis),
   3. advanced arteriosclerotic disease or complicated diabetes mellitus,
   4. chronic obstructive pulmonary disease (COPD) requiring oxygen therapy,
   5. acute or progressive hepatic disease,
   6. acute or progressive renal disease,
   7. congestive heart failure
5. surgery planned during the study period
6. bleeding diathesis
7. history of hypersensitivity to any component of the study medication or chemically related substances
8. history of any anaphylaxis, serious vaccine reactions, or allergy to any of the vaccine component
9. known or suspected impairment/alteration of immune function, for example resulting from:

   1. receipt of immunosuppressive therapy (any corticosteroid therapy or cancer chemotherapy),
   2. receipt of immunostimulants,
   3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within 3 months prior to Visit 1 or planned during the full length of the study,
   4. high risk for developing an immunocompromising disease
10. history of drug or alcohol abuse
11. laboratory-confirmed influenza disease within 6 months prior to Visit 1
12. receipt of influenza vaccine within 6 months prior to Visit 1
13. receipt of another vaccine within 60 days prior to Visit 1, or planned vaccination within 3 weeks following study vaccination
14. any acute respiratory disease or infections requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) or experienced fever (i.e., axillary temperature ≥ 38 degree C) within 5 days prior to Visit 1
15. if female, pregnant or breastfeeding
16. if female, refusal to use a reliable contraceptive method during the three weeks following vaccination
17. planned relocation abroad during the study period
18. any condition that, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2005-09; Primary Completion 2005-10 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines & Diagnostics
Locations (2):
- Lithuania (2):
  - 2nd Department of Internal Diseases, Panevezys Hospital,, Panevezys
  - Dept. Infectious Diseases and Microbiology of Vilnius University, Vilnius

REFERENCES:
- [Result] Ambrozaitis A, Groth N, Bugarini R, Sparacio V, Podda A, Lattanzi M. A novel mammalian cell-culture technique for consistent production of a well-tolerated and immunogenic trivalent subunit influenza vaccine. Vaccine. 2009 Oct 9;27(43):6022-9. doi: 10.1016/j.vaccine.2009.07.083. Epub 2009 Aug 8. PMID 19666152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1200 subjects were enrolled from 2 sites in Lithuania. Of the 1200 subjects enrolled, 700 (58%) were randomized in site 1 and 500 (42%) in site 2. Baseline characteristics, outcome measures, and adverse event summary are based on retrospective analysis which excluded data from site 2.
Pre-assignment Details: All participants enrolled were included in the trial.
Groups:
- cTIV (Combined): Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine from one of three vaccine Lots (Lot1, Lot2 or Lot3).
- TIV Group: Subjects in this group received one dose of Egg derived Trivalent Subunit Influenza Vaccine (TIV).
Period: Overall Study
Arm/Group | cTIV (Combined) | TIV Group
Started | 1029 | 171
Completed | 1024 | 171
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: 1200 subjects were enrolled from 2 sites in Lithuania. Of the 1200 subjects enrolled, 700 (58%) were randomized in site 1 and 500 (42%) in site 2. Baseline characteristics, outcome measures, and adverse event summary are based on retrospective analysis which excluded data from site 2, and include 700 subjects: 600 cTIV, 100 TIV
Groups:
- Total: Total of all reporting groups
Arm/Group | cTIV (Combined) | TIV Group | Total
Number analyzed (Participants) | 600 | 100 | 700
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (11.1) | 26.9 (11.5) | 27.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 321 | 58 | 379
  Male | 279 | 42 | 321
Region of Enrollment [Number; unit: participants]
  Lithuania | 600 | 100 | 700

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine in Adult Subjects
Description: The haemagglutinin Inhibition (HI) antibody titer response following
  1. one dose of cTIV for each of the three lots separately and
  2. one dose of cTIV (combined) compared to TIV is reported as Geometric mean titers (GMTs).
  The HI GMTs were evaluated using egg-derived antigen assay.
Time Frame: Day 22 postvaccination
Population: This analysis was done on per protocol (PP) population defined as all subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol deviation.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- cTIV_lot1: Subjects in this group received one dose of Cell-Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 1.
- cTIV_lot 2: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 2
- cTIV_lot3: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 3.
Arm/Group | cTIV_lot1 | cTIV_lot 2 | cTIV_lot3 | cTIV (Combined) | TIV Group
Number analyzed (Participants) | 198 | 193 | 198 | 589 | 98
Titers
  A/H3N2 strain (day 1) | 12 [11 to 14] | 15 [13 to 17] | 16 [14 to 19] | 14 [13 to 16] | 15 [12 to 18]
  A/H3N2 strain (day 22) | 175 [147 to 207] | 171 [144 to 203] | 158 [133 to 188] | 168 [152 to 185] | 186 [146 to 236]
  A/H1N1 strain (day 1) | 20 [17 to 24] | 20 [17 to 25] | 21 [17 to 25] | 20 [18 to 22] | 22 [18 to 29]
  A/H1N1 strain (day 22) | 390 [326 to 466] | 364 [303 to 436] | 366 [306 to 437] | 373 [335 to 415] | 329 [253 to 428]
  B strain (day 1) | 13 [11 to 15] | 17 [14 to 19] | 14 [12 to 16] | 14 [13 to 16] | 16 [13 to 20]
  B strain (day 22) | 131 [113 to 151] | 157 [136 to 182] | 128 [111 to 148] | 138 [126 to 151] | 124 [99 to 154]

2. Primary Outcome: Geometric Mean Ratios After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine in Adult Subjects
Description: Immunogenicity was assessed in terms of Geometric Mean Ratio (GMR) following
  1. one dose of cTIV for each of the three vaccine lots separately and
  2. for one dose of cTIV (combined) compared to TIV, according to the CHMP criterion.
  The European licensure (CHMP) criterion is met if the mean geometric increase (GMR, day 22/day 1) in HI antibody titer is >2.5.
Time Frame: Day 22 postvaccination
Population: The analysis was performed as PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- cTIV_lot1: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 1.
- TIV Group: Subjects in this group received one dose of Egg-Derived Trivalent Subunit Influenza Vaccine(TIV).
Arm/Group | cTIV_lot1 | cTIV_lot 2 | cTIV_lot3 | cTIV (Combined) | TIV Group
Number analyzed (Participants) | 198 | 193 | 198 | 589 | 98
Ratio
  A/H1N1 strain (Day22/Day1) | 20 [16 to 24] | 18 [14 to 22] | 18 [14 to 22] | 18 [16 to 21] | 15 [11 to 20]
  A/H3N2 strain (Day22/Day1) | 14 [12 to 17] | 11 [9.55 to 14] | 9.92 [8.28 to 12] | 12 [11 to 13] | 12 [9.57 to 16]
  B strain (Day22/Day1) | 10 [8.59 to 12] | 9.42 [7.97 to 11] | 9.37 [7.94 to 11] | 9.63 [8.71 to 11] | 7.53 [5.88 to 9.65]

3. Primary Outcome: Percentage of Subjects With HI Titers ≥40
Description: Immunogenicity was assessed in terms of percentage of adult subjects achieving HI titers ≥40, after
  1. one dose of cTIV for each of the three vaccine lots separately and
  2. for one dose of cTIV (combined) compared to TIV, according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving HI titers ≥40 is >70%.
Time Frame: Day 22 postvaccination
Population: This analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages
Groups:
- cTIV_lot 1: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 1.
- cTIV_lot 3: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 3.
Arm/Group | cTIV_lot 1 | cTIV_lot 2 | cTIV_lot 3 | cTIV (Combined) | TIV Group
Number analyzed (Participants) | 198 | 193 | 198 | 589 | 98
Percentages
  A/H1N1 strain (day 1) | 36 [29 to 43] | 38 [31 to 46] | 34 [27 to 41] | 36 [32 to 40] | 38 [28 to 48]
  A/H1N1 strain (day 22) | 97 [94 to 99] | 97 [93 to 99] | 94 [90 to 97] | 96 [94 to 98] | 97 [91 to 99]
  A/H3N2 strain (day 1) | 19 [14 to 25] | 31 [24 to 38] | 28 [22 to 35] | 26 [22 to 30] | 28 [19 to 37]
  A/H3N2 strain (day 22) | 92 [88 to 96] | 93 [88 to 96] | 91 [86 to 95] | 92 [90 to 94] | 97 [91 to 99]
  B strain (day 1) | 25 [19 to 32] | 31 [25 to 38] | 25 [19 to 31] | 27 [23 to 31] | 31 [22 to 41]
  B strain (day 22) | 92 [88 to 96] | 94 [90 to 97] | 93 [89 to 96] | 93 [91 to 95] | 93 [86 to 97]

4. Primary Outcome: Percentage of Subjects With Seroconversion or Significant Increase in HI Antibody Titers After One Dose of Either Cell-derived or Egg-derived Subunit Trivalent Influenza Vaccine
Description: Immunogenicity was assessed in terms of percentage of adult subjects showing seroconversion or significant increase in HI antibody titers after
  1. one dose of cTIV for each of the three vaccine lots separately and
  2. one dose of cTIV (combined) compared to TIV, according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving seroconversion or significant increase is >40%.
  As per European Licensure (CHMP) criterion seroconversion is defined as percentage of subjects with a prevaccination HI titer <10 to a postvaccination titer ≥40; whereas, significant increase is defined as HI titer ≥10 prevaccination and ≥4-fold Hi titer increase post-vaccination.
Time Frame: Day 22 postvaccination
Population: This analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | cTIV_lot1 | cTIV_lot 2 | cTIV_lot3 | cTIV (Combined) | TIV Group
Number analyzed (Participants) | 198 | 193 | 198 | 589 | 98
Percentages
  A/H1N1 strain | 80 [74 to 86] | 81 [75 to 86] | 82 [76 to 87] | 81 [78 to 84] | 76 [66 to 84]
  A/H3N2 strain | 84 [78 to 89] | 79 [72 to 84] | 78 [71 to 83] | 80 [77 to 83] | 88 [80 to 94]
  B strain | 79 [72 to 84] | 81 [75 to 87] | 80 [74 to 85] | 80 [77 to 83] | 70 [60 to 79]

5. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine.
Description: To assess the safety and tolerability in terms of number of subjects reporting solicited adverse events following one injection of
  1. one dose of cTIV for each of the three vaccine lots separately and
  2. for one dose of cTIV (combined) compared to TIV.
Time Frame: Day 1 to Day 7 postvaccination
Population: Analysis was done on safety dataset.
Measure: Number; unit: subjects
Groups:
- cTIV_lot2: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine (cTIV) from Lot 2.
Arm/Group | cTIV_lot1 | cTIV_lot2 | cTIV_lot3 | cTIV (Combined) | TIV Group
Number analyzed (Participants) | 200 | 199 | 200 | 599 | 100
subjects
  Any Local | 57 | 40 | 37 | 134 | 16
  Injection site ecchymosis | 6 | 7 | 3 | 16 | 5
  Injection site erythema | 32 | 18 | 16 | 66 | 8
  Injection site induration | 11 | 13 | 6 | 30 | 6
  Injection site swelling | 10 | 7 | 6 | 23 | 4
  Injection site pain | 33 | 23 | 24 | 80 | 10
  Any Systemic | 62 | 53 | 55 | 170 | 29
  Chills | 18 | 13 | 10 | 41 | 9
  Malaise | 36 | 29 | 26 | 91 | 15
  Myalgia | 14 | 13 | 11 | 38 | 8
  Arthralgia | 6 | 8 | 5 | 19 | 2
  Headache | 32 | 31 | 31 | 94 | 16
  Sweat | 8 | 15 | 11 | 34 | 4
  Fatigue | 39 | 29 | 32 | 100 | 17
  Fever (>=38C) | 1 | 1 | 2 | 4 | 1
  Other | 13 | 3 | 15 | 31 | 9
  Stayed home due to reaction | 7 | 3 | 7 | 17 | 3
  Analgesic Antipyretic medication used | 10 | 2 | 10 | 22 | 8

6. Secondary Outcome: Safety Data of Subjects Upto Six Months After One Dose of Cell Culture Derived or Egg-derived Influenza Vaccine
Description: Additional safety data from day 1 through day 181 after one dose of cTIV (combined) or TIV in terms of serious adverse events (SAEs), adverse events (AEs) necessitating a physician's visit and/or resulting in premature subject's withdrawal from study is reported.
Time Frame: Day 1 - Day 181 postvaccination
Population: This analysis was done on safety dataset.
Measure: Number; unit: subjects
Groups:
- cTIV (Combined) Day 1 to Day 22: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine from one of three vaccine Lots (Lot 1, Lot2 or Lot3).
- cTIV (Combined) Day 23 to Day 181: Subjects in this group received one dose of Cell Derived Trivalent Subunit Influenza Vaccine from one of three vaccine Lots (Lot1, Lot2 or Lot3).
- TIV Group Day 1 to Day 22; TIV Group Day 23 to Day 181: Subjects in this group received one dose of Egg Derived Trivalent Subunit Influenza Vaccine (TIV).
Arm/Group | cTIV (Combined) Day 1 to Day 22 | cTIV (Combined) Day 23 to Day 181 | TIV Group Day 1 to Day 22 | TIV Group Day 23 to Day 181
Number analyzed (Participants) | 599 | 571 | 100 | 97
subjects
  Any AEs | 74 | 62 | 13 | 6
  At least possibly related AEs | 45 | 1 | 10 | 0
  Serious AEs | 2 | 14 | 0 | 2
  At least possibly related SAEs | 0 | 0 | 0 | 0
  Death | 0 | 1 | 0 | 0
  AE leading to withdrawal | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through out the study period
Description: Postinjection solicited AE were collected from Day1-7. Other AE's and SAEs were collected through out the study period (Day 1 to 6 months).
  Overall, 1200 subjects were enrolled from 2 sites. AE event summary are based on retrospective analysis which excluded data from site 2, and include 700 subjects: 600 cTIV, 100 TIV.
  In cTIV group, 599/600 subjects were included in safety dataset as one subject did not receive the vaccination and withdrew on Day 1.
Arm/Group | cTIV (Combined) | TIV Group
Serious Adverse Events (participants affected / at risk) | 16/599 | 2/100
Other Adverse Events (participants affected / at risk) | 237/599 | 35/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (Combined) (N=599) | TIV Group (N=100)
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 4 | 1
Rhinitis (Infections and infestations) | 1 | 0
Injury Asphyxiation (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Schizoid Personality Disorder (Psychiatric disorders) | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0
Essential Hypertension (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (Combined) (N=599) | TIV Group (N=100)
Chills (General disorders) | 41 | 9
Fatigue (General disorders) | 100 | 17
Injection Site Erythema (General disorders) | 66 | 8
Injection Site Induration (General disorders) | 30 | 6
Injection Site Pain (General disorders) | 80 | 10
Malaise (General disorders) | 92 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 8
Headache (Nervous system disorders) | 95 | 16
Rhinitis (Infections and infestations) | 19 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 34 | 4

LIMITATIONS AND CAVEATS:
Because of potential issues related to Good Clinical Practice (GCP), data from one of the sites were not used in the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days